CLINICAL TRIAL: NCT06694480
Title: A First-in-Human Phase 1 Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of FID-022 as Monotherapy in Patients With Advanced Solid Tumors
Brief Title: Study of FID-022 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fulgent Pharma LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FID-022-001
Record Dates: First submitted 2024-11-12; First posted 2024-11-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: FID-022 treatment Single arm study with 6 planned dose levels.
  Intravenous Administration of FID-022, infusion on day 1 and 8 of each 21-day cycle:
  Dose level 1: 20 mg/m2. Dose level 2: 40 mg/m2. Dose level 3: 60 mg/m2. Dose level 4: 80 mg/m2. Dose level 5: 100 mg/m2. Dose level 6: 120 mg/m2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation (Experimental): Patients will be sequentially enrolled at progressively higher dose levels to receive FID-022 as monotherapy. According to the study design, maintaining the dose level or moving down a dose level will possibly happen when conditions are met.
  Intravenous Administration of FID-022, infusion on day 1 and 8 of each 21-day cycle:
  Dose level 1: 20 mg/m2. Dose level 2: 40 mg/m2. Dose level 3: 60 mg/m2. Dose level 4: 80 mg/m2. Dose level 5: 100 mg/m2. Dose level 6: 120 mg/m2.
  Interventions: Drug: FID-022

INTERVENTIONS:
Drug: FID-022 — Advanced solid tumors

SUMMARY:
The goal of this Phase I Clinical Trial is to evaluate the safety and tolerability of FID-022 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
FID-022-001 is a Phase 1, multicenter, open label dose escalation clinical study of FID-022 as monotherapy. FID-022 is composed of topoisomerase inhibitors encapsulated with a polyethyloxazoline material. The study drug is administered through intravenous route. Patients with advanced solid tumor diagnosis without standard curative treatments are the target population (please see the eligibility section)

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to provide informed consent before the start of any study-specific procedures.
2. Age ≥18 years old.
3. Histologically- or cytologically confirmed malignant solid tumor that is metastatic, unresectable, progressive, or recurrent, and for which there are no standard curative measures, or for whom irinotecan is considered an appropriate palliative treatment option. Patients with known primary brain tumors will be excluded.
4. Measurable disease according to RECIST version 1.1.
5. Adequate treatment washout period of ≥21 days or 5 half-lives, whichever is shorter, for prior chemotherapy, radiotherapy, hormonal therapy, biological therapy, or immunotherapy before the first infusion of FID-022. Note: Palliative radiation is permitted but not ≤14 days before the first infusion of FID-022.
6. ECOG PS of 0 or 1.
7. Recovery from any toxic effects of previous chemotherapy, immunotherapy, targeted therapy, or radiotherapy, as judged by the investigator, to Grade ≤1 according to NCI-CTCAE version 5.0 with the following exceptions: alopecia any grade; and adequately controlled anorexia, fatigue, peripheral neuropathy, or hypothyroidism that must have recovered to Grade ≤2.
8. Adequate bone marrow and organ function defined as the following and these criteria need to be met:

   Bone marrow function
   * ANC ≥1500/mm3 [growth factor administration is not permitted ≤2 weeks from cycle 1 day 1 (C1D1)]
   * Platelet count ≥100,000/mm3 (platelet transfusion is not permitted ≤2 weeks from C1D1)
   * Hemoglobin ≥10 g/dL (criteria must be met without packed red blood cell transfusion ≤2 weeks from C1D1; chronic treatment with erythropoietin is permitted if the patient is on erythropoietin for ≥8 weeks)

   Blood clotting function

   • International normalized ratio (INR) ≤1.5 × upper limit of normal (ULN) and activated partial thromboplastin time ≤1.5 × ULN (except patients who are receiving therapeutic anticoagulation and whose INR should be within the therapeutic range)

   Renal function

   • Measured or Calculated creatinine clearance (using the Cockcroft Gault formula) ≥60 mL/min.

   Hepatic function
   * Normal bilirubin or ≤1.0 mg/dL if the local ULN is less than 1.0 mg/dL.
   * For patients with confirmed liver metastasis, total bilirubin within 1.5 x ULN limit is allowed.
   * Both aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × ULN or ≤5 × ULN if liver metastases present
9. An estimated life expectancy of at least 3 months based on investigator judgment.
10. Male patients and female patients of childbearing potential must agree to use 2 highly effective methods of contraception or practice abstinence from 2 weeks before the first FID-022 infusion and throughout the study. After receiving the last FID-022 dose, female and male patients must agree to continue with 2 highly effective methods for at least 6 and 3 months, respectively. Male patients must refrain from donating sperm during the same period.
11. Negative serum pregnancy test result at screening and on Cycle 1 Day 1 for female patients of childbearing potential.
12. Female patients who are not of childbearing potential should meet at least 1 of the following criteria: have undergone a documented hysterectomy and/or bilateral oophorectomy; have medically confirmed ovarian failure, or achieved postmenopausal status (defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause, or have a serum follicle stimulating hormone level within the laboratory's reference range for postmenopausal women).

Exclusion Criteria:

1. Known hypersensitivity to irinotecan (also called camptothecin-11 [CPT-11]) and/or similar compounds (e.g., topotecan, Trodelvy®).
2. History of any secondary malignancy, with the exception of non-melanoma skin cancers and in situ cancers (such as the following: bladder, gastric, colon, cervical/dysplasia, melanoma, prostate, or breast), or has undergone potentially curative therapy with no evidence of disease recurrence for at least 2 years before the first FID-022 infusion and no additional therapy will be required during the study.
3. Patients with known symptomatic active brain metastases, gliomas, leptomeningeal carcinomatosis, or spinal cord compression or other primary brain tumors. Patients with adequately treated and asymptomatic brain metastases are eligible to participate in the study. Asymptomatic brain metastases are defined as having no neurological symptoms for at least 4 weeks before the first FID-022 infusion without evidence of radiographic progression after treatment, no requirements for corticosteroids within 7 days of the first FID-022 infusion, and no lesion ≥1.5 cm at time of screening. Patients with asymptomatic brain metastases may participate but will require regular imaging of the brain as a site of disease.
4. Received >3 prior lines of chemotherapy for recurrent or metastatic disease unless otherwise discussed with the sponsor's medical monitor or delegate. Chemotherapy given as part of treatment for locally advanced disease in the adjuvant or neoadjuvant setting is not considered a line of prior therapy for recurrent/metastatic disease if completed at least 6 months before the start of FID-022. Similarly, treatment with targeted agents or biologic agents such as naked antibodies as single agents or maintenance treatments will not count as a line of chemotherapy. Antibody drug conjugates are considered as lines of chemotherapy.
5. Medical history of interstitial pulmonary disease, intestinal obstructions, intestinal inflammatory disease and gastrointestinal bleeding, especially those developed from prior irinotecan treatments may not be enrolled.
6. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders that, in the judgment of the investigator, could compromise the patient's safety or the study data integrity.
7. Known history of uncontrolled HIV infection defined as CD4+ cells <350/mm3.
8. Patients with a positive viral load assay at time of screening for hepatitis C or hepatitis B. Patients with adequately treated viral hepatitis and a negative viral load assay are permitted.
9. Requirement of systemic steroids at daily doses >10 mg prednisone equivalent systemic exposure daily, including for control of symptoms.
10. Use of any UDP glucuronosyltransferase family 1 member A1 (UGT1A1) or cytochrome P450 3A4 (CYP3A4) inhibitor or UGT1A1 or CYP3A4 inducer in the previous 14 days before the first FID-022 infusion.
11. Patients with known UGT1A1 deficiency including Gilbert's syndrome (GS).
12. QTcF≥ 470 msec, as calculated by Fridericia formula.
13. Current or recent participation in a study of an investigational product in the prior 4 weeks. Note: Patients who have completed the treatment phase of an investigational study and have entered the follow-up phase of the investigational study may participate in FID-022-001 as long as it has been ≥4 weeks before the first FID-022 infusion.
14. Pregnancy, breastfeeding, or plans to become pregnant during the study or within 24 weeks after the last FID-022 infusion.
15. Plans to donate/bank or retrieve eggs (ova, oocytes) during the study or within 24 weeks after the last FID-022 infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
MTD determination | Through study completion, approximately 2.5 years
  Determine the Maximum Tolerated Dose (MTD) of FID-022 in patients with advanced solid tumors
Number of participants with a treatment-related adverse events as assessed by NCI-CTCAE version 5.0. | Through study completion, approximately 2.5 years
  Frequency and severity of abnormal clinical laboratory results, adverse events (AEs), severity of serious AEs (SAEs) and deaths graded according to the NCI-CTCAE version 5.0
Number of Participants with Dose Limiting Toxicity (DLT) events during the DLT monitoring period (first 21 days of dosing) | 21 days
  DLTs graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5 .0. Maximum tolerated dose (MTD) will be determined based on DLT per protocol.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters: Maximum observed plasma concentration (Cmax) of FID-022 and its components, major metabolites | Up to Day 22
  Identify the peak plasma concentration Cmax for 1). FID-022 as the original drug, 2). released two active components and 3). major known metabolites.
Pharmacokinetic (PK) parameters: Time to the maximum observed plasma concentration (Tmax) of FID-022 and its components, major metabolites | Up to Day 22
  Determine time to the maximum observed plasma concentration (Tmax) for 1). FID-022 as the original drug, 2). released two active components and 3). major known metabolites.
Pharmacokinetic (PK) parameters: Area under the plasma concentration time curve (AUC0-t) of FID-022 and its components, major metabolites | Up to Day 22
  Calculated area under the plasma concentration time curve (AUC0-t) of FID-022 with a focus on the key active component.
Pharmacokinetic (PK) parameters: Area under the plasma concentration time curve (AUC0-∞) of FID-022 and its components, major metabolites | Up to Day 22
  Calculated area under the plasma concentration time curve (AUC0-∞) of FID-022 with a focus on the key active component.
Tumor Response Assessment: Objective Response Rate (ORR) determined by the Investigator | Through study completion, approximately 2.5 years
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Tumor Response Assessment: Disease control rate (DCR) determined by the Investigator | Through study completion, approximately 2.5 years
  DCR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) or a stable disease (SD) for at least 4 weeks or longer based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Tumor Response Assessment: Duration of response (DOR) | Through study completion, approximately 2.5 years
  Duration of overall response is defined as the time from the date of first documented CR or PR, assessed by investigator and based on RECIST v. 1.1, to the documented date of progressive disease (PD) or death, whichever occurred first.
Tumor Response Assessment: Time to Response (TTR) | Through study completion, approximately 2.5 years
  TTR is defined as the time from the initial dosing to the date of first documented response to the treatment, e.g. complete response or partial response, assessed by investigator and based on RECIST v. 1.1.
Tumor Response Assessment: Progression free survival (PFS) | Through study completion, approximately 2.5 years
  PFS defined as the time from the date the participant started study drug to the date the participant experiences an event of radiographic disease progression, clinical progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sites, Principal Investigator — Fulgent Pharma LLC.
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No